CLINICAL TRIAL: NCT05777863
Title: The Effects of a Multidomain Lifestyle Intervention on Brain Functioning and Its Relation With Immunometabolic Markers in Ageing: the HELI Study
Brief Title: The Effects of a Multidomain Lifestyle Intervention on Brain Functioning and Its Relation With Immunometabolic Markers in Ageing
Acronym: HELI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Donders Centre for Cognitive Neuroimaging (Other)
Collaborators: Wageningen University and Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3033003.01
Record Dates: First submitted 2022-09-27; First posted 2023-03-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Life Style; Risk Reduction; Cognitive Decline; Aging
MeSH Terms: conditions — Risk Reduction Behavior; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Multidomain lifestyle intervention. Participants are randomized in a 1:1 ratio to a multidomain lifestyle intervention characterized by group-sessions and supervision (high-intensity intervention group) versus access to general lifestyle-related health information in the form of biweekly leaflets which are provided through e-mail (low-intensity intervention group).
Who Masked: Outcomes Assessor
Masking Description: Participants come for baseline outcome measurement visits in Nijmegen and Wageningen prior to randomization. The follow-up measurements are carried out by researchers, investigators and research-assistants who are not guiding the intervention groups, have no contact with included participants after randomization, and are not involved in the randomization process.
  Participants are aware of their group allocation, as it is clear to participants multiple groups are formed which differ in the way the intervention material is provided.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity group (Experimental): The high-intensity group receives a supervised multidomain lifestyle intervention consisting of weekly group meetings. During the weekly group meetings, information and exercises are provided, and participants are able to exchange experiences and advice with other group members.
  Interventions: Behavioral: Multidomain lifestyle intervention
- Low-intensity group (No Intervention): The low-intensity group only receives access to general lifestyle-related health information through biweekly leaflets, which are provided through e-mail.

INTERVENTIONS:
Behavioral: Multidomain lifestyle intervention — A multidomain lifestyle intervention including the following lifestyle domains: (1) diet, (2) physical activity, (3) sleep, (4) stress/mindfulness, and (5) cognitive training.
  Arms: High-intensity group

SUMMARY:
HELI is a multicenter, randomised controlled trial in two Dutch research centres (Donders Centre for Cognitive Neuroimaging, Nijmegen, and the department of Human Nutrition & Health at Wageningen University) among 104 older adults aged 60-75 years who are at risk for cognitive decline with an intervention duration of 26 weeks (roughly 6 months). Participants are randomized in a 1:1 ratio to a multidomain lifestyle intervention characterized by group-sessions and guidance (high-intensity intervention group) versus online access to general lifestyle-related health information in the form of biweekly leaflets (low-intensity intervention group).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent;
* Age between 60-75 years (at pre-screening);
* Fluency in Dutch (speaking, reading and writing);
* Lives near study centres in Nijmegen and Wageningen (max. 50 kilometers of travelling, to ensure study centre visits are possible without excessive travel burden);
* Presence of ≥2 self-reported risk factors for cognitive decline (BMI of 30 or higher, physical inactivity according to World Health Organization guidelines, hypertension [not using hypertensive drugs counts as an additional risk factor], hypercholesterolemia, diabetes type-II, non-symptomatic cardiovascular disease).

Exclusion Criteria:

* Concurrent participation in other intervention trials;
* Technologically illiterate (complete incompetence in working with computers, apps, online questionnaires, etc.);
* No internet access from home;
* Clinical diagnosis of ≥1 of the following: vascular event (CVA), neurological pathology (e.g. mild cognitive impairment, dementia, multiple sclerosis, Parkinson's, epilepsy), current malignant disease(s) (with or without current treatment), current psychiatric disorder(s) (e.g. depression, psychosis, bipolar episodes), symptomatic cardiovascular disease (e.g. stroke, angina pectoris, heart failure, myocardial infarction), revascularisation surgery in the last 12 months at pre-screening, inflammatory bowel disease (characterised with diarrhoea), visual impairment (e.g. blindness), hearing or communicative impairment;
* Unable to undergo MRI (e.g. metal objects in upper body, past brain surgery, active implants, claustrophobic);
* Cognitive impairment as determined by the Telephone Interview for Cognitive Status (TICS-M1), performed during pre-screening before inclusion.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Change in brain activity during working memory | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Blood-oxygen level dependent activity during N-back (2-back) fMRI task
Change in working memory performance | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Task accuracy during N-back (2-back) fMRI task
Change in cerebral perfusion levels | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Cerebral perfusion measured using arterial spin labelling (ASL)
Change in inflammatory profile in blood plasma: hs-CRP | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Blood plasma inflammatory profile analysis to measure hs-CRP level
Change in inflammatory profile in blood plasma: IL-6 | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Blood plasma inflammatory profile analysis to measure IL-6 level
Change in inflammatory profile in blood plasma: TNF-α | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Blood plasma inflammatory profile analysis to measure TNF-α level
Change in microbiota profile | Change between Baseline (T0) and Follow-up after 6 months (T1)
  16S rRNA based profile of gut microbiota in faeces

SECONDARY OUTCOMES:
Change in Body mass index | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Measured in kg/m^2
Change in Waist circumference | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Measured in cm
Change in Hip circumference | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Measured in cm
Change in Blood pressure | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Measured by blood pressure monitor. Scores range from approximately (for diastolic) 60-120 and (for systolic) 100-180 mmHg, with higher scores indicating higher blood pressure.
Change in Abdominal fat distribution (neuroimaging) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Visceral adipose tissue(VAT)/subcutaneous adipose tissue (SAT) ratio measured by abdominal T1-weighted MRI scan
Change in Brain structure volume profile (neuroimaging) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Brain structure volumes (grey matter, white matter, brain vesicles), measured by MP2RAGE structural sequence
Change in Brain myo-inositol levels (neuroimaging) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Brain myo-inositol levels reflecting local neuroinflammation in dorsolateral prefrontal cortex and hippocampus, measured by magnetic resonance spectroscopy (MRS)
Intracranial iron deposition (neuroimaging) | Baseline (T0)
  Local aggregation of iron deposition within the brain, measured by quantitative susceptibility mapping (QSM)
Change in Neuropsychological test battery scoring | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Z-scoring of cognitive assessments targeting cognitive domains predominantly affected by cognitive ageing: executive function (incl. working memory), episodic memory and processing speed
Change in Trail Making Test A (TMT-A) Numbers : trial time (cognitive assessment) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Discrete number; score 0 - no maximum (seconds to assessment completion). Lower score indicates a better outcome
Change in Trail Making Test A (TMT-A) Numbers: errors (cognitive assessment) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Discrete number; score 0 - no maximum (amount of errors). Lower score indicates a better outcome
Change in Trail Making Test B (TMT-B) Numbers and Letters : trial time (cognitive assessment) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Discrete number; score 0 - no maximum (seconds to assessment completion). Lower score indicates a better outcome
Change in Trail Making Test B (TMT-B) Numbers and Letters: errors (cognitive assessment) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Discrete number; score 0 - no maximum (amount of errors). Lower score indicates a better outcome
Change in Verbal Fluency Test (VFT) (cognitive assessment) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Word count in one minute; score 0 - no maximum. Higher score indicates a better outcome
Change in Rey Auditory Verbal Learning Test (RAVLT): learning trials (cognitive assessment) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Discrete number; score 0 - 15 (amount of words remembered during learning trial 1 to 5). Higher score indicates a better score
Change in Rey Auditory Verbal Learning Test (RAVLT): delayed recall (cognitive assessment) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Discrete number; score 0 - 15 (amount of words remembered during delayed recall). Higher score indicates a better score
Change in Digit Symbol Substitution Test (DSST) (cognitive assessment) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Discrete number; score 0 - 90 (amount of symbols correctly substituted). Higher score indicates better outcome
Change in Wechsler Adult Intelligence Scale (WAIS) digit span (cognitive assessment) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Discrete number; score 0 - 90 (amount of digit spans correctly repeated). Higher score indicates better outcome
Change in Five Facet Mindfulness Questionnaire (questionnaire) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Self-assessment of mindfulness; score 24 - 120. Higher score indicate more mindfulness
Change in Sedentary Behaviour Questionnaire (questionnaire) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Average hours and minutes of sedentary behavior a day; score 0 - 24 hours. Higher score (more hours) indicates more sedentary behavior
Change in Eetscore food questionnaire (questionnaire) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Dutch Healthy Diet Index 2015; score 0 - 160. Higher score indicates a better outcome
Change in Perceived Stress Scale (questionnaire) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Stress perception; score 0 - 40. Higher score indicate more perceived stress
Change in Pittsburgh Sleep Quality Index (PSQI) (questionnaire) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Sleep quality; score 0 - 21. Higher score (referred to as global or total score) indicates worse sleep quality
Change in SQUASH (questionnaire) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Physical activity. METs derived from the Ainsworth's compendium of physical activity will be used to classify physical activity intensity (<1.5METs- sedentary, 1.6-2.9 METs- light, 3.0-5.9METs- moderate, >6.0- vigorous physical activity)
Change in Cognitive Failures Questionnaire (questionnaire) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Subjective cognitive functioning; score 0 - 100. A higher score indicates more subjective cognitive failure
Change in Memory Self-Efficacy MIA (questionnaire) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Self-evaluation and confidence of memory. Sum of Part 1 + Part 2A and B. Part 1: Strategy (scores 10 - 50, higher scores indicate more use of strategies), Part 2A: Subjective memory functioning (score 23 - 115, higher score indicates better memory self-efficacy) and Part 2B: Locus (score 7 - 35, higher scores indicate better perceived personal control over remembering abilities)
Change in total amount of bacteria, fungi and specific bacterial strains (faeces) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Total amount of bacteria, fungi and specific bacterial strains are quantified using digital droplet PCR in faecal samples
Change in individual short-chain fatty acids (SCFAs) profile (faeces) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  GC-MS and LC-MS measurements to assess profile of individual SCFAs in faecal samples (acetic acid, formic acid, propionic acid, isobutyric acid, butyric acid, isovaleric acid, valeric acid, 4-methyl valeric acid, hexanoic acid, heptanoic acid)
Change in microbiome-derived bioactive compounds (faeces) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Amount of microbiome-derived bioactive compounds is measured by untargeted LC-MS microbiota-derived metabolite analysis in faecal samples
Change in intestinal inflammation profile (faeces) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Assay-based profile of intestinal inflammation measured in faecal samples
Change in Gut transit time | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Gut transit time measured by blue muffin consumption and appearance in faeces
Change in metabolic profile (blood) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Assay-based profile of (energy) metabolism measured in plasma samples
Change in inflammation profile (blood) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Assay-based profile of systemic inflammation measured in plasma samples
Change in intestinal integrity profile (blood) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Assay-based profile of intestinal integrity measured in plasma samples
Change in brain health profile (blood) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Assay-based profile of brain health measured in plasma samples
Change in white blood cell count (blood) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  White blood cell count measured via finger prick analysis
Change in small intestinal bacterial overgrowth (SIBO) (breath) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Measurement of total exhaled hydrogen gas after glucose consumption in breath samples

OTHER OUTCOMES:
Montreal Cognitive Assessment (MOCA) (cognitive assessment) | Baseline (T0)
  Discrete number; score 0 - 30. Higher score indicates better cognitive performance (≥26 indicates normal cognitive functioning)
Baseline Demographics and medical history (questionnaire) | Baseline (T0)
  Demographic information, medical history and medication use - qualitative assessment
Change in 4DKL (questionnaire) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  (Psychosocial) complaints in daily life; separate scores for distress (>10 moderate, >20 severe), depression (>2 moderate, >5 severe), anxiety (>3 moderate, >9 severe) and somatisation (>10 moderate, >20 severe)
Change in EQ-5D-5L (questionnaire) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Quality of life; score 0 - 100. Higher score indicate better quality of life
Change in LIBRA (questionnaire) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Modifiable dementia risk using lifestyle for brain health; score -5.9 - +12.7. Higher score indicates a worse outcome (higher dementia risk)
Change in Lubben Social Network Scale (questionnaire) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Social contact and perceived social support; score 0 - 30. Higher score indicates a better outcome (higher level of perceived social support)
Change in SARC-F Sarcopenia questionnaire (questionnaire) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Sarcopenia; score 0 - 10 (i.e. 0-2 points for each component; 0 = best to 10 = worst)
Change in Cognitive Emotions Regulation Questionnaire (questionnaire) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Cognitive coping strategies. Answers are scored on a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree). The scoring takes the average of all the scores in each subscale of cognitive reappraisal and expressive suppression
Change in Hospital Anxiety and Depression Scale (questionnaire) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Anxiety and depression; separate scores for anxiety (0 - 21) and depression (0 - 21). For each domain, a score >8 indicates psychiatric condition of anxiety or depression
Change in Starkstein Apathy Scale (questionnaire) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Screen and measure apathetic symptoms. A higher total score (range 0-42) indicates more severe apathy, with a score greater than 14 or greater is indicative of clinical apathy
Change in COVID status (questionnaire) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Vaccination status, COVID history - qualitative assessment
Change in Gastrointestinal symptoms questionnaire (questionnaire) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Gastrointestinal symptoms, qualitative assessment
Change in Bristol stool chart (questionnaire) | Change between Baseline (T0) and Follow-up after 6 months (T1)
  Classification of faeces type, qualitative assessment

CONTACTS AND LOCATIONS:
Overall Officials: Esther Aarts, PhD, Principal Investigator — Donders Centre for Cognitive Neuroimaging
Locations (2):
- Netherlands (2):
  - Donders Centre for Cognitive Neuroimaging, Nijmegen, Gelderland
  - Wageningen University & Research, Wageningen, Gelderland